CLINICAL TRIAL: NCT00996502
Title: A Phase I/II Study of Bevacizumab and Erlotinib in Combination With Docetaxel and Prednisone for Patients With Hormone Refractory Prostate Cancer
Brief Title: Study of Bevacizumab and Erlotinib for Patients With Hormone Refractory Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor enrollment; PI left the institution
Sponsor: Columbia University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB8399
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Bevacizumab; Erlotinib Hydrochloride; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination regimen (Experimental): Bevacizumab, Erlotinib, Docetaxel, Prednisone (dose escalation)
  Phase I:
  * Cohort 1: 55mg/m2 of Docetaxel on Day 1 of the cycle, 15mg/kg of Bevacizumab every 3 weeks, 200 mg of Erlotinib PO daily days 2-16, 5 mg of Prednisone PO bid
  * Cohort 2: 65mg/m2 of Docetaxel on Day 1 of the cycle, 15mg/kg of Bevacizumab every 3 weeks, 200 mg of Erlotinib PO daily days 2-16, 5 mg of Prednisone PO bid
  * Cohort 3: 75mg/m2 of Docetaxel on Day 1 of the cycle, 15mg/kg of Bevacizumab every 3 weeks, 200 mg of Erlotinib PO daily days 2-16, 5 mg of Prednisone PO bid
  Interventions: Drug: Docetaxel; Drug: Bevacizumab; Drug: Erlotinib; Drug: Prednisone

INTERVENTIONS:
Drug: Docetaxel — Phase I:
  * Cohort 1: 55mg/m2 of Docetaxel on Day 1 of the cycle
  * Cohort 2: 65mg/m2 of Docetaxel on Day 1 of the cycle
  * Cohort 3: 75mg/m2 of Docetaxel on Day 1 of the cycle
  Other Names: Taxotere
Drug: Bevacizumab — 15mg/kg of Bevacizumab every 3 weeks
  Other Names: Avastin
Drug: Erlotinib — 200 mg of Erlotinib PO daily days 2-16
  Other Names: Tarceva
Drug: Prednisone — 5 mg of Prednisone PO bid
  Other Names: Prednicot

SUMMARY:
The primary objectives of this study are to evaluate the safety and best dose of a regimen including bevacizumab and erlotinib in combination with docetaxel and prednisone. In addition, the investigators wish to evaluate how well these drugs might work against this disease. Bevacizumab and erlotinib are novel drugs that attack the blood vessels supplying the tumor cells and attack a receptor on the tumor cells, respectively. This study has two parts. In the first part of the study, eighteen patients will be enrolled. Patients will receive escalating doses of docetaxel in combination with standard doses of bevacizumab and erlotinib until the safest dose is determined. An additional 37 patients will enter into the second part of the study and all will receive the safest dose. In this part of the study, the effectiveness of this regimen against hormone refractory prostate cancer (HRPC) will be monitored by evaluating prostate-specific antigen (PSA) and objective response of the tumor.

DETAILED DESCRIPTION:
In this Phase I/Phase II study, the primary objectives are to establish the maximum tolerated dose of docetaxel, erlotinib, bevacizumab, and prednisone in patients with metastatic hormone refractory prostate cancer and to determine the efficacy of this regimen for treatment of metastatic HRPC. In the phase I portion of the study, eligible patients will be enrolled and treated using a "3+3" design. Docetaxel will be started at 55 mg/m2 every cycle (21 days) and dose escalated by 10 mg/m2 at each cohort level. The dose of bevacizumab will be held constant at 15 mg/kg every 3 weeks and erlotinib will be provided at 200 mg PO daily from days 216 as described in previous safety studies. All patients will receive prednisone 5 mg PO bid. Eighteen patients will be treated in the phase I portion. The phase II dose for this combined treatment will be defined as either the highest dosage cohort in which 6 patients are treated and there are less than 3 dose limiting toxicities (DLTs); or the combination of docetaxel, erlotinib, and bevacizumab at the cohort 3 dose level, whichever is the lower dose. Another 37 patients will be enrolled for the phase II study. All patients will receive the phase II recommended dose as determined by the phase I portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented diagnosis of prostate adenocarcinoma (PCa) not amenable to curative therapy.
* Evidence of progressive metastatic disease.
* Surgically or medically castrated. Patients must continue on medical castration (LHRH agonists) throughout protocol participation. Patients who have discontinued LHRH agonists should be restarted on therapy. Testosterone levels should be obtained prior to protocol initiation and should be less than 50 ng/mL.
* Previous antiandrogen and hormonal therapies must have been discontinued prior to protocol initiation.
* Receiving bisphosphonate therapies should have had this therapy started at least 4 weeks prior to treatment initiation and should be on a stable dose. Although being on bisphosphonate therapy is not an exclusion to the study, bisphosphonate therapy should not be started during the study.
* Fully recovered and greater than 4 weeks from any major surgery or radiation therapy. There must be greater than 8 weeks from last dose of radionucleotide administration. There must be greater than 7 days from minor surgical procedures (eg portacath insertion, fine needle aspirations or core biopsies).
* No previous cytotoxic therapy including estramustine or suramin. No previous therapies with anti-angiogenic agents including thalidomide or bevacizumab.
* No history of brain metastases.
* No current congestive heart failure (defined as New York Heart Association Class II, III, or IV).
* Well-controlled blood pressure. Those with a history of hypertension should be well-controlled on a regimen of anti-hypertensive medication (exclude if BP>150/100).
* No history of significant bleeding (e.g. upper or lower gastrointestinal bleeding or hemoptysis) within 6 months of protocol enrollment.
* No history of gastrointestinal perforation, intraabdominal fistula, or intraabdominal abscess within 6 months of protocol enrollment.
* No history of arterial thrombotic events within 6 months of protocol enrollment.
* No active serious non-healing wound, ulcer, or bone fracture.
* Eastern Cooperative Oncology Group (ECOG) performance status between 0 and 1.
* > 18 years old.
* Adequate hematopoietic and organ function.
* Able to swallow capsules.
* Willing to use effective means of contraception for study duration and for at least 3 months after the completion of protocol therapy.
* Able to provide informed consent.

Exclusion Criteria:

* Active second malignancy other than basal or squamous skin cancer. Patients who have completed all necessary therapy and are considered to have less than a 30% risk of relapse by their physician are not thought to have an active second malignancy.
* Serious concurrent uncontrolled medical disorder.
* Disease for whom corticosteroids are contraindicated such as an active peptic ulcer or uncontrolled diabetes. Patients with controlled diabetes may be considered but must be made aware that their diabetic medications may require adjustment.
* Received prior treatment with a tyrosine kinase inhibitor, estimated glomerular filtration rate inhibitor (EGFR), or vascular endothelial growth factor (VEGF) inhibitor. For the phase II trial, patients who have had previous cytotoxic therapy will not be eligible.
* Currently or have recently participated in a clinical trial (within 4 weeks from the first day of treatment) or are receiving investigational therapies.
* Unable to comply with study or follow-up procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Petrylak, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to the IRB in March 2010.
Groups:
- Combination Regimen: Bevacizumab, Erlotinib, Docetaxel, Prednisone (dose escalation)
  Phase I:
  * Cohort 1: 55mg/m2 of Docetaxel on Day 1 of the cycle, 15mg/kg of Bevacizumab every 3 weeks, 200 mg of Erlotinib PO daily days 2-16, 5 mg of Prednisone PO bid
  * Cohort 2: 65mg/m2 of Docetaxel on Day 1 of the cycle, 15mg/kg of Bevacizumab every 3 weeks, 200 mg of Erlotinib PO daily days 2-16, 5 mg of Prednisone PO bid
  * Cohort 3: 75mg/m2 of Docetaxel on Day 1 of the cycle, 15mg/kg of Bevacizumab every 3 weeks, 200 mg of Erlotinib PO daily days 2-16, 5 mg of Prednisone PO bid
  Docetaxel: Phase I:
  * Cohort 1: 55mg/m2 of Docetaxel on Day 1 of the cycle
  * Cohort 2: 65mg/m2 of Docetaxel on Day 1 of the cycle
  * Cohort 3: 75mg/m2 of Docetaxel on Day 1 of the cycle
  Bevacizumab: 15mg/kg of Bevacizumab every 3 weeks
  Erlotinib: 200 mg of Erlotinib PO daily days 2-16
  Prednisone: 5 mg of Prednisone PO bid
Period: Overall Study
Arm/Group | Combination Regimen
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combination Regimen
Number analyzed (Participants) | 4
Age, Customized [Number; unit: participants]
  18 years and older | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Docetaxel in Combination With Erlotinib, Bevacizumab, and Prednisone (Phase I)
Time Frame: After three 21-day cycles
Population: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in March 2010.
Arm/Group | Combination Regimen
Number analyzed (Participants) | 0

2. Secondary Outcome: Objective Response Rate at the Recommended Phase II Dose Level of Docetaxel, Bevacizumab, Erlotinib, and Prednisone
Time Frame: Every 9 weeks
Population: as for outcome 1
Arm/Group | Combination Regimen
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival Rate
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Combination Regimen
Number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Patients Alive at One Year (Phase II)
Time Frame: One year
Population: as for outcome 1
Arm/Group | Combination Regimen
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the AE data.
Arm/Group | Combination Regimen
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No